CLINICAL TRIAL: NCT04651322
Title: Quantified Analysis of Neuronal Recovery Using Myelin Imaging After Robot Assisted Upper Arm Training in Subacute Stroke Patients: Randomized Controlled Trial
Brief Title: Quantified Analysis of Neuronal Recovery Using Myelin Imaging After Robot Assisted Upper Arm Training in Subacute Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2019-0023
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental)
  Interventions: Device: upper robot Robot assisted upper arm training(RAT)
- Control group (Other)
  Interventions: Behavioral: Conventional therapy

INTERVENTIONS:
Device: upper robot Robot assisted upper arm training(RAT) — The training group received an additional upper robot Robot assisted upper arm training(RAT) with Armeopower® 5 times per week for 4weeks.
  *Robot Assisted Arm training + Conventional occupational therapy
  Arms: Training group
Behavioral: Conventional therapy — The control group received the usual conventional therapy *Only Conventional occupational therapy
  Arms: Control group

SUMMARY:
* Quantitative assessment method developed for brain plasticity through disability rehabilitation using a brain imaging technique.
* Development of brain imaging technology to improve understanding of brain plasticity during rehabilitation and to improve the efficiency of rehabilitation treatment for people with brain injury. ○ Development of the latest brain function image analysis algorithm and data processing technology

  * Development of new technology for imaging brain plasticity in addition to existing functional imaging technology and diffuse imaging technology (Example: Myelinated brain imaging technology, susceptibility imaging (SWI) technology)
  * Development of image reconstruction software technology using new image technology
  * Multi-image and repeated shot data processing technology, wheat analysis technology development (Example: 3D registration technology, automated segmentation technology)
* Conducted clinical research on clinical quantitative evaluation of brain plasticity due to rehabilitation treatment

  * Recruitment of a group of patients for pursuing plasticity through rehabilitation among stroke patients (estimating the number of sample patients by setting a specific patient group and analyzing statistical power)
  * Image-based brain change analysis through patient rehabilitation and before and after imaging
  * Comparative analysis through securing a control group and activating the control group. Derivation of clinical relevance through comparison with rehabilitation process

ELIGIBILITY:
Inclusion Criteria:

1. less than 6 months after onset of the stroke
2. have FMA score greater than 7
3. have confirmed that the integrity of the Corticospinal Tract (CST) is preserved in Diffusion Tensor Imaging (DTI) taken using
4. over 20 years of age
5. can understand and participated in study
6. consented to this study in writing or verbally

Exclusion Criteria:

1. quadriplegia
2. past history of stroke
3. past history of Musculoskeletal disease or history of Neurological diseases
4. have a history of injury to the upper limb and upper chest, surgery, or peripheral nerve damage
5. have skin ulcers or skin diseases such as open wounds that have difficulty applying RAT
6. Pregnant woman
7. If it is judged that this clinical participation is not appropriate according to the judgment of medical doctor

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | before training(0week)
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia
Fugl-Meyer Assessment (FMA) | after training(4week)
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia

CONTACTS AND LOCATIONS:
Overall Officials: Deog Young Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No